CLINICAL TRIAL: NCT01868945
Title: Dose Finding Study in Physically Frail Elderly to Measure 25(OH) Vitamin D Levels After Supplementation With Hy.D Calcifediol 25 SD/S and Vitamin D3
Acronym: D-DOSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2012-10-24-HyD
Record Dates: First submitted 2013-05-24; First posted 2013-06-05 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Pre-frail Elderly; Frail Elderly
Keywords: Vitamin D3; Calcifediol 25; Frail; Dose-response
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5 µg/day Hy.D Calcifediol (Experimental)
  Interventions: Dietary Supplement: 5 µg/day Hy.D Calcifediol
- 10 µg/day Hy.D Calcifediol (Experimental)
  Interventions: Dietary Supplement: 10 µg/day Hy.D Calcifediol
- 15 µg/day Hy.D Calcifediol (Experimental)
  Interventions: Dietary Supplement: 15 µg/day Hy.D Calcifediol
- 20 µg/day vitamin D3 (Active Comparator)
  Interventions: Dietary Supplement: 20 µg/day vitamin D3

INTERVENTIONS:
Dietary Supplement: 5 µg/day Hy.D Calcifediol — 5 µg/day Hy.D Calcifediol taken together with breakfast for a total period of 24 weeks
  Arms: 5 µg/day Hy.D Calcifediol
Dietary Supplement: 10 µg/day Hy.D Calcifediol — 10 µg/day Hy.D Calcifediol taken together with breakfast for a total period of 24 weeks
  Arms: 10 µg/day Hy.D Calcifediol
Dietary Supplement: 15 µg/day Hy.D Calcifediol — 15 µg/day Hy.D Calcifediol taken together with breakfast for a total period of 24 weeks
  Arms: 15 µg/day Hy.D Calcifediol
Dietary Supplement: 20 µg/day vitamin D3 — 20 µg/day vitamin D3 taken together with breakfast for a total period of 24 weeks
  Arms: 20 µg/day vitamin D3

SUMMARY:
The purpose of this study is to assess the dose of Hy.D Calcifediol 25 SD/S (a metabolite of vitamin D3) which will achieve the range of mean serum 25(OH)D between 75-100nmol/L in physically frail elderly people after 24 weeks of daily supplementation with different doses of Hy.D Calcifediol 25 SD/S compared to vitamin D3.

ELIGIBILITY:
Inclusion Criteria:

* 25(OH)D levels between 25 - 50 nmol/L;
* Age 65 and older;
* Physically frail, based on the criteria designed by Fried et al. [1]. Frailty will be defined as a clinical syndrome in which one or more of the following criteria are present: unintentional weight loss (4.5 kg in past year), selfreported exhaustion (CES-D questionnaire), weakness (grip strength), slow walking speed and low physical activity (Minnesota questionnaire). These criteria are easily assessable and have been commonly used to determine frailty;
* Men and women;
* Body mass index between 20 and 35 kg/m2 (used for stratification);
* Willingness and ability to comply with the protocol.

Exclusion Criteria:

* Medical Illness: malabsorption syndrome: known intestinal malabsorption, celiac diseases, inflammatory bowel disease; diseases that may enhance serum calcium concentration: sarcoidosis, lymphoma, kidney stone in the last 10 years, primary hyperparathyroidism; abnormal indices of calcium metabolism, uncontrolled hypocalcaemia; diagnosed renal insufficiency, diagnosed cancer, diagnosed liver failure.
* Hypercalcemia : serum calcium adjusted for albumin of > 2.6 nmol/L.
* Medication: bisphosphonate or Parathyroid hormone (PTH) treatment, tuberculostatics, epilepsy medication, interfering with vitamin D metabolism and vitamin D supplementation.
* Use of vitamin D supplementation in the last three months (excluding multivitamin supplementation).
* Not willing to stop the use of multivitamin supplementation during the study.
* (Expected) increase in exposure to sunlight (e.g. travelling to a sunny resort).
* Patient heavily consumes alcohol containing products defined as greater than (>) 3 drinks (beer, wine, or distilled spirits) of alcoholic beverages per day.
* Donating blood in the period of 2 months before, until 1 month after the end of the study.
* Planned surgery.
* Participation in another clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mean serum 25(OH)D levels in Hy.D and vitamin D3 supplemented groups at baseline | Baseline (day 0)
  Outcome measurement: Mean serum 25(OH)D levels at baseline before supplementation of three doses of Hy.D and 1 dose of vitamin D3.
Mean serum 25(OH)D levels in Hy.D and vitamin D3 supplemented groups after 4 weeks | 4 weeks after initial compound intake
  Outcome measurement: Mean serum 25(OH)D levels after 4 weeks of supplementation of three doses of Hy.D and 1 dose of vitamin D3.
Mean serum 25(OH)D levels in Hy.D and vitamin D3 supplemented groups after 8 weeks | 8 weeks after initial compound intake
  Outcome measurement: Mean serum 25(OH)D levels after 8 weeks of supplementation of three doses of Hy.D and 1 dose of vitamin D3.
Mean serum 25(OH)D levels in Hy.D and vitamin D3 supplemented groups after 12 weeks | 12 weeks after initial compound intake
  Outcome measurement: Mean serum 25(OH)D levels after 12 weeks of supplementation of three doses of Hy.D and 1 dose of vitamin D3.
Mean serum 25(OH)D levels in Hy.D and vitamin D3 supplemented groups after 16 weeks | 16 weeks after initial compound intake
  Outcome measurement: Mean serum 25(OH)D levels after 16 weeks of supplementation of three doses of Hy.D and 1 dose of vitamin D3.
Mean serum 25(OH)D levels in Hy.D and vitamin D3 supplemented groups after 20 weeks | 20 weeks after initial compound intake
  Outcome measurement: Mean serum 25(OH)D levels after 20 weeks of supplementation of three doses of Hy.D and 1 dose of vitamin D3.
Mean serum 25(OH)D levels in Hy.D and vitamin D3 supplemented groups after 24 weeks | 24 weeks after initial compound intake
  Outcome measurement: Mean serum 25(OH)D levels after 24 weeks of supplementation of three doses of Hy.D and 1 dose of vitamin D3.

SECONDARY OUTCOMES:
Descriptive: 25(OH)D3 serum steady state reached? | 0, 4, 8, 12, 16, 20, 24 weeks after study start
  Assessment if 25(OH)D3 serum levels will reach a steady state after 24 weeks supplementation of 3 doses of Hy.D and 1 dose of vitamin D3

CONTACTS AND LOCATIONS:
Overall Officials: Lisette De Groot, Prof, Principal Investigator — Wageningen University; Michael Tieland, PhD, Principal Investigator — Wageningen University; Luc van Loon, Prof, Principal Investigator — Maastricht University
Locations (1):
- Wageningen University, Wageningen, Wageningen, Netherlands

REFERENCES:
- [Derived] Vaes AMM, Tieland M, de Regt MF, Wittwer J, van Loon LJC, de Groot LCPGM. Dose-response effects of supplementation with calcifediol on serum 25-hydroxyvitamin D status and its metabolites: A randomized controlled trial in older adults. Clin Nutr. 2018 Jun;37(3):808-814. doi: 10.1016/j.clnu.2017.03.029. Epub 2017 Mar 31. PMID 28433267